CLINICAL TRIAL: NCT02688959
Title: A Feasibility/Pilot Trial of a Motor Attention Training Intervention for College Students With ADHD
Brief Title: Motor Attention Training for Attention Deficit Hyperactivity Disorder (ADHD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-0807; A348700 (Other: UW Madison); VCRGE\WAISMAN CENTER\WAISMAN (Other: UW Madison); Protocol version 15 July 2024 (Other: IRB UW, Madison)
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: motor attention training; exercise; tai chi; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity | interventions — Tai Ji; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tai Chi (Experimental): Participants in this arm will attend 50-minute classes 2 times per week for 8 weeks. The course will emphasize experiential learning with 2 weeks of introductory sessions on gait, posture, and tai chi principles followed by instruction in the 24-form Yang style sequence. Students will be given a video to aid learning outside of class, and maintenance of practice post-intervention.
  Interventions: Behavioral: Tai Chi
- Exercise (Active Comparator): Participants in the exercise arm will attend 50-minute classes 2 times per week for 8 weeks. The course will emphasize cardio-aerobic fitness training. Students will be given a video to aid practice outside of class, and maintenance of practice post-intervention.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Participants in the control arm will not attend a class and not be given a video.

INTERVENTIONS:
Behavioral: Tai Chi
  Arms: Tai Chi
Behavioral: Exercise
  Arms: Exercise

SUMMARY:
The investigators will perform a feasibility/pilot trial of two non-pharmacological interventions for ADHD in college students.

DETAILED DESCRIPTION:
College students diagnosed with ADHD will be randomized to three arms of approximately 8 weeks duration: (1) standard care plus a tai chi class, (2) standard care plus an exercise class, and (3) standard care alone. The exercise class will control for the social and motor components of tai chi training. The investigators will determine methodological parameters relevant to a subsequent full scale trial including recruitment and retention rates, acceptance of randomization, adherence to the interventions, and variance in outcome measures. The primary clinical outcome measure of this pilot randomized controlled trial (RCT) will be pre- to post-intervention change in inattention, i.e. the Inattentive Symptoms subscale of the Conners Adult ADHD Rating Scale self-report long form (CAARS-S:L, see Interviews etc. "Converse_S_L"). Secondary measures to be explored will include self- and informant-report, neurocognitive measures, psychophysiological measures, and academic performance. Practice time will be assessed daily and follow-up self-report of ADHD symptoms will be gathered monthly for 3 months beyond the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* University of Wisconsin-Madison enrolled undergraduate
* Documented ADHD diagnosis

Exclusion Criteria:

* Unable or unwilling to participate in the interventions

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Estimated)
Dates: Start 2016-02; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms of inattention | 8 weeks
  Inattentive Symptoms subscale of the Conners Adult ADHD Rating Scale self-report long form (CAARS-S:L). The total range of scores is 0-27 with higher scores indicating more severe symptom levels.

SECONDARY OUTCOMES:
Feasibility of implementing wireless Electroencephalogram(EEG) to measure the theta beta ratio during performance of tai chi. | up to 90 minute
  Feasibility of implementing wireless EEG will be assessed by the quality of EEG data. Acceptable data should have satisfactory signal to noise characteristics. Satisfactory signal to noise ratio will be evaluated by the variance within individual across trials of the ratio of occipital alpha power between the eyes closed and eyes open conditions. Feasibility will be judged by the criterion that the coefficient of variance (CV = s.d./mean) be less than 1/3.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander K Converse, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Waisman Center, Madison, Wisconsin, United States

REFERENCES:
- [Background] Converse AK, Ahlers EO, Travers BG, Davidson RJ. Tai chi training reduces self-report of inattention in healthy young adults. Front Hum Neurosci. 2014 Jan 27;8:13. doi: 10.3389/fnhum.2014.00013. eCollection 2014. PMID 24478679
- [Result] Converse AK, Barrett BP, Chewning BA, Wayne PM. Tai Chi training for attention deficit hyperactivity disorder: A feasibility trial in college students. Complement Ther Med. 2020 Sep;53:102538. doi: 10.1016/j.ctim.2020.102538. Epub 2020 Aug 14. PMID 33066865
- See also: Converse personal site — http://brainimaging.waisman.wisc.edu/~converse/